CLINICAL TRIAL: NCT00058656
Title: A Phase I/II Study of Xcellerated T Cells(tm) in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Autologous T Cell Immunotherapy for Chronic Lymphocytic Leukemia (CLL) Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xcyte Therapies (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT004
Record Dates: First submitted 2003-04-08; First posted 2003-04-10 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2005-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Immunotherapy; T Cell Therapy; Adoptive immunotherapy; Xcellerate; Xcellerated
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

INTERVENTIONS:
Procedure: Infusion of Activated & Expanded Autologous T Cells

SUMMARY:
Patients will have immune cells collected and then expanded outside of the body. Patients will receive an infusion of a large number of expanded immune cells. There will be three dose levels studied. The goal of the study will be to determine the safety as well as potential efficacy of this treatment.

DETAILED DESCRIPTION:
This is a Phase I/II single arm dose escalation study of a novel T cell immunotherapy for chronic lymphocytic leukemia (CLL). Patients will receive one dose of Xcellerated T Cells(tm), an ex vivo activated and expanded autologous T cell product, in an attempt to enhance immune responses with anti-tumor activity. This study is being conducted to test the safety and determine the maximum tolerated dose (MTD) of Xcellerated T Cells in patients with CLL. In addition, lymphocyte counts, lymph node area, and quantitative immunoglobulins will be assessed for preliminary evidence of a therapeutic effect. In correlative studies, changes in the phenotype of T and B lymphocytes will be evaluated by flow cytometry. Changes in T cell repertoire and anti-tumor immune activity will also be assessed. It is expected that 12 to 18 patients will be treated.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of CLL at any time in the past, as defined by all of the following:

> 5 x 109 peripheral blood lymphocytes/L which are positive for CD5 and one or more B cell markers (CD19, CD20, CD23).

< 55% of lymphocytes identified as prolymphocytes

* Intermediate or High Risk disease as defined by the Modified 3-stage system
* Patients with Intermediate Risk (Rai Stages I and II) must have active disease, as determined by one or more of the following criteria:

  1. One or more of the following disease related symptoms i. Weight loss > 10% within the previous 6 months ii. Fevers of greater than 100.5°F for > 2 weeks iii. Night sweats without evidence of infection
  2. Massive (i.e. > 6 cm below the left costal margin) or progressive splenomegaly
  3. Massive lymph nodes or clusters (i.e. > 10 cm in longest diameter) or progressive lymphadenopathy
  4. Progressive lymphocytosis with an increase of >50% over a 2-month period, or an anticipated doubling time of less than 12 months
* T cells (CD3+) comprising > 1.5% and < 10 % of peripheral white blood cells as assessed by flow cytometry
* CD4+/CD8+ of > 0.30, as assessed by flow cytometry
* Age of at least 18 years
* ECOG performance status of 0 to 2
* Life expectancy 6 months
* Able to comprehend and provide signed informed consent
* Women of childbearing potential must have a negative serum pregnancy test and agree to use a medically accepted form of contraception from the time of initial screening through completion of the study

Exclusion Criteria

* Evidence of Richter's Syndrome, T cell CLL, prolymphocytic leukemia, hairy-cell leukemia, splenic lymphoma with villous lymphocytes, large granular lymphocytosis, Sezary-cell leukemia, adult T-cell leukemia/lymphoma, or leukemic manifestations of non-Hodgkin's lymphoma
* Receipt of any chemotherapy, monoclonal antibody, investigational, or other systemic therapy for the treatment of CLL within 2 months prior to registration.
* Receipt of glucocorticoids (with the exception of inhaled glucocorticoid steroids for the use of allergic rhinitis or pulmonary disease) within 2 months prior to registration
* Receipt of intravenous immunoglobulin (IVIG) within 1 month of registration
* Registration for, or plans to participate in, any other clinical trial concurrently for the duration of this trial
* History of malignancy other than CLL within five years of registration, except adequately treated basal or squamous cell skin cancer or in situ carcinoma of the cervix. Other exceptions must be approved by the Xcyte Therapies' Medical Monitor prior to registration.
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within seven days of registration
* Liver disease or hepatitis as reflected by a serum bilirubin or ALT > 2.0 times the upper limit of normal laboratory range within 15 days of registration
* Compromised renal function as reflected by a serum creatinine > 2 times the upper limit of normal laboratory range within 15 days of registration
* History of autoimmune disease unrelated to CLL (e.g., rheumatoid arthritis, multiple sclerosis, systemic lupus erythematosis). Autoimmune disease related to CLL, e.g. idiopathic thrombocytopenic purpura (ITP) or autoimmune hemolytic anemia, is permitted if treatment with steroids has not been required in the two months prior to registration. Hypothyroidism without evidence of Grave's Disease or Hashimoto's thyroiditis is permitted.
* Major organ system dysfunction including (but not limited to): New York Heart Association Class III or IV (Appendix B, page 51), pulmonary disease requiring the use of inhaled steroids or bronchodilators, renal, hepatic, gastrointestinal, neurologic, or psychiatric dysfunction which would impair patient's ability to participate in the trial
* Evidence of infection with HIV 1 or 2, HTLV 1 or 2
* Evidence of acute or active chronic Hepatitis B or C infection
* Positive human anti-mouse antibody (HAMA) test as performed at the central reference laboratory designated by the sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-03

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frohlich, MD, Study Director — Xcyte Therapies
Locations (4):
- United States (4):
  - University of California, San Diego, San Diego, California
  - Atlanta Cancer Care, Roswell, Georgia
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - MD Anderson Cancer Center, Houston, Texas